CLINICAL TRIAL: NCT03038607
Title: Effect of Low-dose Aspirin on Fetal Weight of Idiopathic Asymmetrically Intrauterine Growth Restricted Fetuses With Abnormal Umbilical Doppler Indices
Brief Title: Aspirin in Asymmetrically Intrauterine Growth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASP
Record Dates: First submitted 2017-01-29; First posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Intrauterine Growth Restriction Asymmetrical
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin group (Active Comparator)
  Interventions: Drug: Aspirin
- No intervention (No Intervention)

INTERVENTIONS:
Drug: Aspirin — This group were subjected to aspirin 75 mg once daily for 6 weeks.
  Arms: Aspirin group

SUMMARY:
Intrauterine growth restriction refers to a fetus that has failed to get a specific measures by a gestational age. Asymmetric type of Intrauterine growth restriction is known by normal sized head with smaller abdomen.It is important to recognize the growth restricted fetuses, because these fetuses may have fetal or neonatal complications.

When blood flow is increased, the oxygen and nutrients will deliver good to the fetus. The role of low-dose aspirin therapy in management of intrauterine growth restriction is controversial. It has been used, in many studies, in prevention of intrauterine growth restriction especially in women at high risk of pre-eclampsia or obstetrical antiphospholipid syndrome.

ELIGIBILITY:
Inclusion Criteria:

* The pregnant women
* 28-30 weeks
* Idiopathic asymmetrically intrauterine growth restriction
* Middle aged women (20-35 years)
* Women with abnormal umbilical artery Doppler flow indices ( > +2 standard deviation above mean for gestational age)

Exclusion Criteria:

* Women less than 20 and more than 35 years
* hypertensive or diabetic women
* any type of smoking
* multiple pregnancies
* amniotic fluid index <5 cm
* premature pre-labor rupture of membranes
* abnormal placenta
* any fetal congenital malformations.
* women had absent diastolic flow or reversed flow in umbilical artery at the time of recruitment.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Estimated fetal weight | 6 weeks

SECONDARY OUTCOMES:
Birth weight | 6 weeks
Changes in Doppler blood flow indices in umbilical artery | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes